CLINICAL TRIAL: NCT02352662
Title: Peri-operative Assessment of Coagulopathy in Neonates and Infants Undergoing Cardiac Surgery
Status: Withdrawn | Type: Observational
Why Stopped: Competition with another study.
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, David Faraoni, Cardiac Anesthesiologist, Boston Children's Hospital
Other Study IDs: IRB-P00016002
Record Dates: First submitted 2015-01-26; First posted 2015-02-02 (Estimated); Last update posted 2017-04-10 (Actual); Status verified 2017-04

CONDITIONS: Congenital Heart Disease
Keywords: Congenital Heart Disease; Point-of-care coagulation monitoring; Rotaional Thromboelastometry
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Collect bloods samples at three different time points intraoperatively to look at coagulation factors
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Study Group: Three blood samples will be collected intra-operatively from each subject enrolled
  Interventions: Other: Perioperative blood samples collection

INTERVENTIONS:
Other: Perioperative blood samples collection — Collect blood samples at 3 different points intra-operatively. Each blood sample will be run using rotational thromboelastometry to assess intraoperative coagulation

SUMMARY:
This prospective study will aim to globally assess the coagulopathy induced during cardiac surgery with cardiopulmonary bypass (CPB) in a large pediatric population. The investigators primary objective will be the understanding of CPB-induced coagulopathy based on demographic and surgical characteristics, and coagulation assays. Secondary objective will aim at determining the relationship between coagulation assays, postoperative blood loss, and transfusion requirements. The ultimate goal will be to design an algorithm using point-of-care monitoring that could be used to guide hemostatic therapies in neonates and children undergoing cardiac surgery.To do this, investigators will examine the coagulation in the laboratory based setting.

ELIGIBILITY:
Inclusion Criteria:

* Neonates weighing greater than 2.5 kg
* Patients equal to or less than 12 months of age
* Undergoing elective cardiac surgery with cardiopulmonary bypass

Exclusion Criteria:

* Emergent procedure
* The patient is deemed to be in a moribund condition (American Society of Anesthesiology (ASA 5))

Max Age: 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Neonates and infants undergoing cardiac surgery with cardiopulmonary bypass
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Evidence of CPB-induced coagulopathy confirmed by coagulation assays | Over 6 months

CONTACTS AND LOCATIONS:
Overall Officials: David Faraoni, MD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Miller BE, Mochizuki T, Levy JH, Bailey JM, Tosone SR, Tam VK, Kanter KR. Predicting and treating coagulopathies after cardiopulmonary bypass in children. Anesth Analg. 1997 Dec;85(6):1196-202. doi: 10.1097/00000539-199712000-00003. PMID 9390579
- [Background] Faraoni D, Willems A, Romlin BS, Belisle S, Van der Linden P. Development of a specific algorithm to guide haemostatic therapy in children undergoing cardiac surgery: a single-centre retrospective study. Eur J Anaesthesiol. 2015 May;32(5):320-9. doi: 10.1097/EJA.0000000000000179. PMID 25387300
- [Background] Paparella D, Brister SJ, Buchanan MR. Coagulation disorders of cardiopulmonary bypass: a review. Intensive Care Med. 2004 Oct;30(10):1873-81. doi: 10.1007/s00134-004-2388-0. Epub 2004 Jul 24. PMID 15278267
- [Background] Arnold P. Treatment and monitoring of coagulation abnormalities in children undergoing heart surgery. Paediatr Anaesth. 2011 May;21(5):494-503. doi: 10.1111/j.1460-9592.2010.03461.x. Epub 2010 Dec 1. PMID 21118327
- [Background] Osthaus WA, Boethig D, Johanning K, Rahe-Meyer N, Theilmeier G, Breymann T, Suempelmann R. Whole blood coagulation measured by modified thrombelastography (ROTEM) is impaired in infants with congenital heart diseases. Blood Coagul Fibrinolysis. 2008 Apr;19(3):220-5. doi: 10.1097/MBC.0b013e3282f54532. PMID 18388502
- [Background] Faraoni D, Savan V, Levy JH, Theusinger OM. Goal-directed coagulation management in the perioperative period of cardiac surgery. J Cardiothorac Vasc Anesth. 2013 Dec;27(6):1347-54. doi: 10.1053/j.jvca.2013.08.005. Epub 2013 Oct 5. No abstract available. PMID 24103717
- [Background] Gorlinger K, Dirkmann D, Hanke AA, Kamler M, Kottenberg E, Thielmann M, Jakob H, Peters J. First-line therapy with coagulation factor concentrates combined with point-of-care coagulation testing is associated with decreased allogeneic blood transfusion in cardiovascular surgery: a retrospective, single-center cohort study. Anesthesiology. 2011 Dec;115(6):1179-91. doi: 10.1097/ALN.0b013e31823497dd. PMID 21970887
- [Background] Williams GD, Bratton SL, Ramamoorthy C. Factors associated with blood loss and blood product transfusions: a multivariate analysis in children after open-heart surgery. Anesth Analg. 1999 Jul;89(1):57-64. doi: 10.1097/00000539-199907000-00011. PMID 10389779
- [Background] Hayashi T, Sakurai Y, Fukuda K, Yada K, Ogiwara K, Matsumoto T, Yoshizawa H, Takahashi Y, Yoshikawa Y, Hayata Y, Taniguchi S, Shima M. Correlations between global clotting function tests, duration of operation, and postoperative chest tube drainage in pediatric cardiac surgery. Paediatr Anaesth. 2011 Aug;21(8):865-71. doi: 10.1111/j.1460-9592.2011.03524.x. Epub 2011 Jan 21. PMID 21251146
- [Background] Jensen AS, Johansson PI, Bochsen L, Idorn L, Sorensen KE, Thilen U, Nagy E, Furenas E, Sondergaard L. Fibrinogen function is impaired in whole blood from patients with cyanotic congenital heart disease. Int J Cardiol. 2013 Sep 1;167(5):2210-4. doi: 10.1016/j.ijcard.2012.06.019. Epub 2012 Jun 22. PMID 22727966
- [Background] Faraoni D, Willems A, Savan V, Demanet H, De Ville A, Van der Linden P. Plasma fibrinogen concentration is correlated with postoperative blood loss in children undergoing cardiac surgery. A retrospective review. Eur J Anaesthesiol. 2014 Jun;31(6):317-26. doi: 10.1097/EJA.0000000000000043. PMID 24503704
- [Background] Faraoni D, Van der Linden P. Factors affecting postoperative blood loss in children undergoing cardiac surgery. J Cardiothorac Surg. 2014 Feb 11;9:32. doi: 10.1186/1749-8090-9-32. PMID 24512988
- [Background] Lacroix J, Hebert PC, Hutchison JS, Hume HA, Tucci M, Ducruet T, Gauvin F, Collet JP, Toledano BJ, Robillard P, Joffe A, Biarent D, Meert K, Peters MJ; TRIPICU Investigators; Canadian Critical Care Trials Group; Pediatric Acute Lung Injury and Sepsis Investigators Network. Transfusion strategies for patients in pediatric intensive care units. N Engl J Med. 2007 Apr 19;356(16):1609-19. doi: 10.1056/NEJMoa066240. PMID 17442904